CLINICAL TRIAL: NCT05197426
Title: A Phase 2, Randomized, Double-Blind, Placebo-controlled Study to Compare Efficacy and Safety of Oral Azacitidine Plus Best Supportive Care Versus Best Supportive Care as Maintenance Therapy in Japanese Subjects With Acute Myeloid Leukemia in Complete Remission
Brief Title: A Study to Compare the Efficacy and Safety of Oral Azacitidine Plus Best Supportive Care Versus Best Supportive Care as Maintenance Therapy in Japanese Participants With Acute Myeloid Leukemia (AML) in Complete Remission
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA055-005
Record Dates: First submitted 2022-01-05; First posted 2022-01-19 (Actual); Results first posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; cc-486

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Oral Azacitidine (Experimental)
  Interventions: Drug: Oral Azacitidine
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Oral Azacitidine — Specified dose on specified days
  Other Names: CC-486; BMS-986345; Onureg
  Arms: Oral Azacitidine
Other: Placebo — Specified dose of specified days
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of oral azacitidine plus best supportive care versus best supportive care as maintenance therapy in a cohort of Japanese participants ≥ 55 years of age with Acute Myeloid Leukemia (AML) and in complete remission/complete remission with incomplete blood count recovery after conventional induction chemotherapy with or without consolidation chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 55 years of age inclusive at the time of signing the informed consent
* Newly diagnosed, histologically confirmed de novo Acute Myeloid Leukemia (AML) or AML secondary to prior myelodysplastic syndrome (MDS) or chronic myelomonocytic leukemia (CMML)
* Should have undergone induction therapy with intensive chemotherapy with or without consolidation therapy as recommended in appropriate guideline(s) or equivalent regimen according to institutional standard: having achieved first complete remission (CR)/complete remission with incomplete blood count recovery (CRi) status within 4 months prior to starting study therapy

Exclusion Criteria:

* Suspected or proven acute promyelocytic leukemia; or AML with previous hematologic disorder such as chronic myeloid leukemia or myeloproliferative neoplasms, excluding MDS and CMML
* Prior bone marrow or stem cell transplantation
* Received therapy with hypomethylating agents for MDS and went on to develop AML within four months of discontinuing the therapy with hypomethylating agents
* Have achieved CR/CRi following therapy with hypomethylating agents

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2026-04-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (31):
- Local Institution - 0011, Huntsville, Alabama, United States
- Japan (30):
  - Local Institution - 0017, Nagoya, Aichi-ken
  - Local Institution - 0023, Nagoya, Aichi-ken
  - Local Institution - 0009, Toyoake, Aichi-ken
  - Local Institution - 0022, Aomori, Aomori
  - Local Institution - 0005, Kamogawa, Chiba
  - Local Institution - 0003, Kashiwa-shi, Chiba
  - Local Institution - 0010, Matsuyama, Ehime
  - Local Institution - 0020, Yoshida Gun, Fukui
  - Local Institution - 0016, Fukuoka, Fukuoka
  - Local Institution - 0014, Ōgaki, Gifu
  - Local Institution - 0001, Maebashi, Gunma
  - Local Institution - 0004, Sapporo, Hokkaido
  - Local Institution - 0019, Kanazawa, Ishikawa-ken
  - Local Institution - 0012, Isehara, Kanagawa
  - Local Institution - 0006, Sagamihara-shi, Kanagawa
  - Local Institution - 0013, Yokohama, Kanagawa
  - Local Institution - 0015, Sendai, Miyagi
  - Local Institution - 0026, Osaka, Osaka
  - Local Institution - 0021, Ōsaka-sayama, Osaka
  - Local Institution - 0031, Shimotsuke, Tochigi
  - Local Institution - 0032, Bunkyo Ku, Tokyo
  - Local Institution - 0002, Shinagawa, Tokyo
  - Local Institution - 0030, Shinjuku-ku, Tokyo
  - Local Institution - 0029, Sumida Ku, Tokyo
  - Local Institution - 0018, Fukuoka
  - Local Institution - 0027, Fukuoka
  - Local Institution - 0008, Nagasaki
  - Local Institution - 0025, Okayama
  - Local Institution - 0028, Saitama
  - Local Institution - 0007, Yamagata

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT05197426.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 19 Participants randomized and treated
Groups:
- Treatment 1: CC-486, 200mg taken for the first 14 days of each 28-day treatment cycle
- Treatment 2: Placebo, 200mg taken for the first 14 days of each 28-day treatment cycle
Period: Treatment
Arm/Group | Treatment 1 | Treatment 2
Started | 12 | 7
Completed (= Ongoing Treatment) | 7 | 1
Not Completed | 5 | 6
Not completed — Disease Relapse | 2 | 2
Not completed — Physician Decision | 1 | 3
Not completed — Transitioned to commercially available treatment | 1 | 0
Not completed — Other Reasons | 1 | 1
Period: Follow Up
Arm/Group | Treatment 1 | Treatment 2
Started | 5 | 6
Completed (= On Going Follow up) | 4 | 3
Not Completed | 1 | 3
Not completed — Death | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment 1 | Treatment 2 | Total
Number analyzed (Participants) | 12 | 7 | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.1 (3.48) | 69.3 (6.85) | 70.4 (4.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 6 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 12 | 7 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 12 | 7 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Recurrence Free Survival (RFS)
Description: The time from randomization to the date of documented relapse after CR or CRi per central review, or death from any cause, whichever occurs first. Participants who are still alive without documented relapse after CR or CRi, or who were lost to follow-up without documented relapse, will be censored at the date of their last response assessment.
Time Frame: Approximately 17.7 months
Population: All Treated Participants
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 12 | 7
Months | NA [10.2 to NA] — Insufficient number of participants with events to calculate via KM methodology | 7.4 [1.4 to NA] — Insufficient number of participants with events to calculate via KM methodology

2. Secondary Outcome: Overall Survival (OS)
Description: The time from randomization to death from any cause and will be calculated using the randomization date and date of death, or date of last follow-up for censored participants. All participants will be followed until dropout, death, or study termination. Participants who dropout or are alive at study termination will have their OS times censored at the time of last contact, as appropriate.
Time Frame: Approximately 17.7 months
Population: All Treated Participants
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 12 | 7
Months | NA [18.1 to NA] — Insufficient number of participants with events to calculate via KM methodology | 15.1 [12.3 to NA] — Insufficient number of participants with events to calculate via KM methodology

3. Secondary Outcome: Time to Relapse From CR or CRi
Description: The interval from the date of randomization to the date of documented relapse after CR or CRi, as defined according to the IWG AML response criteria. Time to relapse will be analyzed using a competing risk analysis where death without documented relapse is treated as a competing risk for relapse from CR/CRi. Similar censoring rules as in primary analysis of RFS will be applied.
Time Frame: Approximately 17.7 months
Population: All Treated Participants
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 12 | 7
Months | NA [10.2 to NA] — Insufficient number of participants with events to calculate via KM methodology | 7.4 [1.4 to NA] — Insufficient number of participants with events to calculate via KM methodology

4. Secondary Outcome: Time to Discontinuation
Description: The interval from the date of randomization to the date of discontinuation from IP. Subjects who are ongoing in treatment at the time of study closure will be censored at the date of last visit.
Time Frame: Approximately 17.7 months
Population: All Treated Participants
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 12 | 7
Months | NA [6.7 to NA] — Insufficient number of participants with events to calculate via KM methodology | 5.8 [1.8 to 10.4]

5. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Time Frame: Approximately 17.7 months
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 12 | 7
Participants
  at least 1 TEAE | 12 | 7
  TEAE related to study drug | 12 | 3
  at least 1 Serious TEAE | 4 | 2
  Serious TEAE releated to study drug | 3 | 1
  Grade 3 or 4 TEAE | 9 | 4
  Grade 3 or 4 TEAE related to study drug | 8 | 1

6. Secondary Outcome: Number of Participants With Clinically Significant Changes in Physical Examination
Description: Number of participants with clinically significant changes in physical examination
Time Frame: Approximately 17.7 months
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 12 | 7
Participants | 0 | 0

7. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Vital signs include the following: systolic blood pressure, diastolic blood pressure, heart rate, respiratory rate, temperature and weight.
Time Frame: Approximately 17.7 months
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 12 | 7
Participants | 0 | 0

8. Secondary Outcome: Number of Participants With Clinically Significant Changes in Clinical Laboratory Examinations
Time Frame: Approximately 17.7 months
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 12 | 7
Participants | 0 | 0

9. Secondary Outcome: Number of Participants Who Received Concomitant Medication
Description: Concomitant medications are defined as non-study medications that are started after the date of randomization but before the end of the study treatment period or started on or before the date of randomization but ended or remain ongoing during the study treatment period.
Time Frame: Approximately 17.7 months
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 12 | 7
Participants | 12 | 7

10. Secondary Outcome: Mean Change From Baseline in Facit-Fatigue Scale
Description: The FACIT-Fatigue Scale is a short, 13-item, easy-to-administer tool that measures an individual's level of fatigue during usual daily activities over the past week. The level of fatigue is measured on a five-point Likert scale (0 = not at all fatigued to 4 = very much fatigued). It has scores that range from 0 to 52, with higher scores indicating less fatigue. Quality of life (QoL)scores on these FACIT scales significantly decline as patient performance status worsens.
Time Frame: From C1D1 to C12D1 (approximately 336 days)
Population: All Treated Participants
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 12 | 7
Score on a Scale
  Cycle 2 Day 1 | 3.2 (6.12) | 2.3 (3.90)
  Cycle 6 Day 1: number analyzed (Participants) | 11 | 4
  Cycle 6 Day 1 | 1.0 (6.94) | -3.0 (8.52)
  Cycle 12 Day 1: number analyzed (Participants) | 9 | 2
  Cycle 12 Day 1 | 3.9 (4.94) | -1.0 (1.41)

11. Secondary Outcome: Mean Change From Baseline in EQ-5D-5L
Description: The European Quality of Life 5D-5L Scale (EQ-5D-5L) assesses general health-related quality of life. Health is defined in 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Responses are coded so that a '1' indicates no problem, and '5' indicates the most serious problem. The responses for the 5 dimensions are combined in a 5-digit number. The EQ-5D-5L health utility index (HUI) is assessed using the Crosswalk algorithm for France based on the individual responses to the 5 EQ-5D-5L domains ranging from -0.530 to 1.000. The smallest change considered clinically meaningful, is defined as a score difference of 0.08 points. The lower the score the better.
Time Frame: From C1D1 to C12D1 (approximately 336 days)
Population: All Treated Participants
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 12 | 7
Score on a Scale
  Cycle 2 Day 1 | 0.0267 (0.12963) | -0.0106 (0.02797)
  Cycle 6 Day 1: number analyzed (Participants) | 11 | 4
  Cycle 6 Day 1 | 0.0413 (0.11735) | -0.0485 (0.23776)
  Cycle 12 Day 1: number analyzed (Participants) | 9 | 2
  Cycle 12 Day 1 | 0.0254 (0.08160) | -0.0855 (0.12092)

12. Secondary Outcome: Pharmacokinetic Evaluation: CMax
Description: Cmax is defined as maximum plasma concentration of the drug.
Time Frame: on C1D1 (after first dose on day 1)
Population: Due to limited data collection only 1 participant had data collected on C1D1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 1 | 0
ng/mL | 155 (NA) — Cannot calculate GCoV with 1 data value. |

13. Secondary Outcome: Pharmacokinetic Evaluation: Tmax
Description: Tmax is defined is the time to maximum plasma concentration
Time Frame: on C1D1 (after first dose on day 1)
Population: Due to limited data collection only 1 participant had data collected on C1D1.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 1 | 0
hours (h) | 0.45 [NA to NA] — Not able to calculate full range with 1 sample collected. |

14. Secondary Outcome: Pharmacokinetic Evaluation: AUC(0-T)
Description: Area under the plasma concentration time-curve. AUC from time 0 to the last time of quantifiable concentration.
Time Frame: on C1D1 (after first dose on day 1)
Population: Due to limited data collection only 1 participant had data collected on C1D1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 1 | 0
h*ng/mL | 284.7 (NA) — Cannot calculate GCoV with 1 data value. |

15. Secondary Outcome: Pharmacokinetic Evaluation: AUC(INF)
Time Frame: on C1D1 (after first dose on day 1)
Population: Due to limited data collection only 1 participant had data collected on C1D1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 1 | 0
h*ng/mL | 287.7 (NA) — Cannot calculate GCoV with 1 data value. |

16. Secondary Outcome: Pharmacokinetic Evaluation: T-Half
Description: the time required for the amount or concentration of a drug to decrease by one-half
Time Frame: on C1D1 (after first dose on day 1)
Population: Due to limited data collection only 1 participant had data collected on C1D1.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 1 | 0
hours (h) | 0.467 [NA to NA] — Not able to calculate full range with 1 sample collected. |

17. Secondary Outcome: Pharmacokinetic Evaluation: CLT/F(INF)
Description: the volume of plasma from which a substance is completely removed per unit time.
Time Frame: on C1D1 (after first dose on day 1)
Population: Due to limited data collection only 1 participant had data collected on C1D1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 1 | 0
mL/min | 11588 (NA) — Cannot calculate GCoV with 1 data value. |

18. Secondary Outcome: Pharmacokinetic Evaluation: Vz/F
Description: the amount of drug in the body to the concentration of drug measured in a biological fluid
Time Frame: on C1D1 (after first dose on day 1)
Population: Due to limited data collection only 1 participant had data collected on C1D1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 1 | 0
mL/min | 469 (NA) — Cannot calculate GCoV with 1 data value. |

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events: (From first dose to last dose + 28 days): Approximately 18.7 months
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Arm/Group | Treatment 1 | Treatment 2
All-Cause Mortality (participants affected / at risk) | 1/12 | 2/7
Serious Adverse Events (participants affected / at risk) | 4/12 | 2/7
Other Adverse Events (participants affected / at risk) | 12/12 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment 1 (N=12) | Treatment 2 (N=7)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment 1 (N=12) | Treatment 2 (N=7)
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 3
Hypoglobulinaemia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 6 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2
Cardiac failure (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 2
Dental caries (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 6 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Trichoglossia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 7 | 1
Chest pain (General disorders) | 1 | 0
Injection site erythema (General disorders) | 0 | 1
Injection site reaction (General disorders) | 1 | 1
Malaise (General disorders) | 1 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0
COVID-19 (Infections and infestations) | 4 | 1
Cystitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Herpes zoster oticus (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Chillblains (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 2 | 2
Tumour marker abnormal (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Sensory disturbance (Nervous system disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 1
Calculus urinary (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-27): https://cdn.clinicaltrials.gov/large-docs/26/NCT05197426/Prot_SAP_000.pdf